CLINICAL TRIAL: NCT03662607
Title: Impact of Virtual Reality on Pre-procedural anxieTy Prior to Heart cathEterIzAtion - VR-THEIA
Acronym: VR-THEIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Ryan Madder, MD, MD, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-074
Record Dates: First submitted 2017-09-27; First posted 2018-09-07 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Preprocedure Anxiety
Keywords: preprocedure; anxiety; cardiac catheterization
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard pre-procedural education for cardiac catheterization.
- Treatment (Experimental): Standard pre-procedural education plus virtual reality experience for cardiac catheterization.
  Interventions: Behavioral: Virtual reality experience

INTERVENTIONS:
Behavioral: Virtual reality experience — * Baseline wellness self-assessment administered (reporting on absence or presence and degree of severity of headache, nausea, dizziness, fatigue and vision abnormalities)
  * Seated comfortably and free of direct obstruction
  * Shown individual components of the VR system (View-Master with smartphone; headphones); given instructions; encouraged to ask questions.
  * Begin the VR experience. Study personnel stay in the room & provide guidance and answer questions regarding the technology
  * When VR experience concluded, wellness self-assessment will be administered again.
  Arms: Treatment

SUMMARY:
The primary aim of this study is to test the hypothesis that use of VR combined with standard procedural education will result in less pre-procedural anxiety than standard procedural education alone among patients undergoing first-time cardiac catheterization. The VR technology being evaluated in this study will allow patients to experience a 3-D simulation of certain aspects of their upcoming procedure prior to the actual procedure date.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a left-heart catheterization procedure at the Meijer Heart Center
* 18-75 years of age
* Signed study consent form

Exclusion Criteria:

* History of cardiac procedure(s) in a cardiac catheterization laboratory
* History of seizures, migraine headaches or severe susceptibility to motion sickness
* Currently taking psychotropic drugs or on long-term psychotropic treatment
* Unable to read and speak English
* Visually impaired
* Unable to provide written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share data at this time.

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Standard preprocedural education
- VR Group (Treatment): Stanard preprocedural education plus viewing of virtual reality video
Period: Overall Study
Arm/Group | Control | VR Group (Treatment)
Started | 91 | 89
Completed | 91 | 89
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients undergoing clinical cardiac catheterization, who voluntarily agreed to study participation
Groups:
- VR Group (Treatment): Standard preprocedural education plus viewing of virtual reality video
- Total: Total of all reporting groups
Arm/Group | Control | VR Group (Treatment) | Total
Number analyzed (Participants) | 91 | 89 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 42 | 88
  >=65 years | 45 | 47 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.52) | 64 (8) | 64 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 65
  Male | 61 | 54 | 115
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 89 | 180

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety Measured by the Sate-Trait Anxiety Inventory (STAI)
Description: The primary outcome of this study is patient anxiety, as measured by the State Trait Anxiety Inventory (STAI) score. STAI is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Time Frame: Change from baseline visit to procedure day. Baseline visits will occur up to 4 weeks prior to procedure.
Measure: Mean (Standard Deviation); unit: Mean STAI score
Arm/Group | Control | VR Group (Treatment)
Number analyzed (Participants) | 91 | 89
Mean STAI score | 69.81 (17.11) | 65.71 (15.22)

ADVERSE EVENTS:
Time Frame: Per patient assigned to the VR arm, baseline assessment was conducted immediately prior to watching the video. The patient was than assessed with the same questionnaire immediately after watching the video. The third and final assessment was conducted 24 hours after watching the video. Therefore, the time frame over which adverse event data were collected was 24 hours.
Description: Monitored VR patients for headache, nausea, dizziness, fatigue, and visual disturbances. Assessments occurred pre-VR viewing, immediate post VR viewing, and 24 hours post procedure.
Groups:
- Treatment: Standard pre-procedural education plus virtual reality experience for cardiac catheterization.
  Virtual reality experience: - Baseline wellness self-assessment administered (reporting on absence or presence and degree of severity of headache, nausea, dizziness, fatigue and vision abnormalities)
  * Seated comfortably and free of direct obstruction
  * Shown individual components of the VR system (View-Master with smartphone; headphones); given instructions; encouraged to ask questions.
  * Begin the VR experience. Study personnel stay in the room & provide guidance and answer questions regarding the technology
  * When VR experience concluded, wellness self-assessment will be administered again.
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/89
Other Adverse Events (participants affected / at risk) | 0/91 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT03662607/Prot_SAP_000.pdf